CLINICAL TRIAL: NCT06366490
Title: Phase 1 Study to Assess the Safety and Immunogenicity of Innocell Autologous Cellular Immunotherapy Administered in Patients With Recurrent Epithelial Ovarian Cancer
Brief Title: Safety and Immunogenicity of Innocell Autologous Cellular Immunotherapy for Recurrent Epithelial Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PhotonPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP2023-001
Record Dates: First submitted 2024-03-28; First posted 2024-04-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer; Recurrent Epithelial Ovarian Cancer Which Includes Epithelial Ovarian, Fallopian Tube and/or Primary Peritoneal Cancer
Keywords: Autologous vaccine; Autologous Cellular Immunotherapy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is a 2-part design. For each participant, Part 1 will involve tissue procurement and confirmation of the ability to manufacture the Innocell vaccine, followed by Part 2 which is the treatment phase, involving Innocell administration to patients.
Masking Description: Open label Phase I trial with no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Innocell an Autologous Cellular Immunotherapy (Experimental): Innocell autologous immunotherapy will be administered with CpG 1018 adjuvant
  Interventions: Biological: Innocell Autologous Cellular Immunotherapy

INTERVENTIONS:
Biological: Innocell Autologous Cellular Immunotherapy — Innocell Autologous Cellular Immunotherapy cells will be administered with CpG 1018 adjuvant ID every 2 weeks x 3 doses

SUMMARY:
Safety and Immunogenicity of Innocell Autologous Cellular Immunotherapy Administered in Patients with Recurrent Epithelial Ovarian Cancer

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-center, pilot study of Innocell autologous cellular immunotherapy (i.e., Innocell vaccine) in patients with recurrent EOC.

The study is a 2-part design. For each participant, Part 1 will involve tissue procurement and confirmation of the ability to manufacture the Innocell vaccine, followed by Part 2 which is the treatment phase, involving Innocell administration to patients.

Part 1 - Tissue Procurement and Manufacturing of Innocell Vaccine

Participants will be screened to assure they fulfill the enrollment criteria. Screening must be performed within 30 days of administration of the Innocell regimen. Patients will undergo biopsy of the tumor. The team will target to harvest 1.0 gram or greater of tissue for the manufacturing process to produce 3 doses of Innocell and overage for testing. Upon successful manufacture and release testing, the Innocell vaccine series will be initiated.

Part 2 - Innocell Administration and Follow-up

Participants will undergo a Baseline Visit to confirm they meet the enrollment criteria. The Baseline Visit must be performed within 14 days of planned initiation of the Innocell vaccine series. The vaccine series will consist of Innocell cells combined with CpG 1018 adjuvant via intradermal (ID) injection every 2 weeks (14 ± 3 days) x 3 doses.

Participants will be monitored for a minimum of 60 minutes following each injection, with a follow up visit 2 days (+2 days) post-each injection for evaluation of safety and tolerability. All participants who received at least 1 dose of Innocell will be followed for safety through a minimum of 30 days after the last dose of Innocell or until all treatment-related adverse events are resolved or returned to Baseline/Grade 1, whichever is longer, or until the Investigator determines the outcome will not change with further followup.

Blood will be drawn for evaluation of immune response and disease burden prior to each dose of Innocell, 2 weeks (+/- 3 days) and 30 (+7) days after the last dose of Innocell.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and female;
2. Has histologically or cytologically confirmed diagnosis of advanced epithelial ovarian cancer (except carcinosarcoma), primary peritoneal, or fallopian tube cancer that has received at least 1 line of platinum-based systemic therapy and for whom single-agent therapy is appropriate as the next line of treatment;
3. Been treated with available standard-of-care therapy likely to convey clinical benefit (i.e., PARP inhibitors for women with germline BRCA mutation and in homologous recombination repair deficiency based on prior molecular testing or bevacizumab as appropriate);
4. Documented relapse or progression on or after the most recent line of therapy;
5. Patients must have at least 2 sites of measurable or detectable disease. The team will target to collect 1.0 gram of tumor tissue that can be removed and be available for manufacturing;
6. Eastern Collaborative Oncology Group (ECOG) performance status (PS) 0-2;
7. Recovery from clinically relevant toxicities to Grade 2 or less (except alopecia, peripheral neuropathy, and ototoxicity);
8. Adequate hematological, hepatic, and renal function obtained ≤ 28 days prior to planned initiation of vaccine series
9. Negative pregnancy test for women of childbearing potential and agree to practice a medically acceptable contraception regimen throughout the participation in the clinical trial; and,
10. Provide written informed consent for study participation.

Exclusion Criteria:

1. Positive clinical history of HIV, HCV, HBV, HTLV-1/2;
2. Diagnosis of immunodeficiency, either primary or acquired;
3. Active or prior history of autoimmune disease;

   Note: The following conditions are permitted (i.e., not exclusionary) if the condition does not require immunosuppressive treatment:
   * Type 1 diabetes (if stable, well controlled, and not brittle); Vitiligo; Hypo- or hyperthyroid disease; or Autoimmune alopecia.
4. Treatment with systemic steroids or any other form of immunosuppressive therapy within 14 days prior to planned initiation of the Innocell vaccine; Note: Inhaled or topical steroids, including mouthwash, and adrenal replacement doses are permitted in the absence of active autoimmune disease.
5. Has any acute infection that requires specific therapy. Acute therapy must be completed at least 7 days prior to initiation of Innocell series;
6. Has received any live or attenuated vaccines against infectious diseases within 28 days of the planned vaccine initiation. Inactive vaccines, including SARS-CoV-2 vaccines authorized for use for active immunization to prevent COVID-19 are allowed and must be given in accordance with the prevailing immunization guidelines; or
7. Has received any other investigational agents within 4 weeks of planned vaccine initiation.
8. Hs received treatment with an approved systemic therapy within 3 weeks of planned vaccine initiation;
9. Prior malignancy, except those that were treated curatively and have not recurred within 5 years prior to study treatment; resected basal cell and squamous cell skin cancers;
10. History or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the patient's participation for the full duration of the study, such that it is not in the best interest of the patient to participate, in the opinion of the treating investigator; or
11. Inability of the subject to comply with study procedures and/or followup.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of autologous manufacturing | 2 months
  Percent success rate to manufacture Innocell from autologous malignant tissue for patient administration
Safety assessed by treatment emergent adverse events | From 1st dose of Innocell until 30 days post last dose
  Proportion of subjects experiencing treatment emergent adverse events

SECONDARY OUTCOMES:
Immune response to Innocell | Baseline to 30 days post last dose of Innocell
  Mean change in circulating biomarkers
Immune response to Innocell | Baseline to 30 days post last dose of Innocell
  Mean change in circulating cytokine levels
Immune response to Innocell | Baseline to 30 days post last dose of Innocell
  Mean change in T-cell counts
Immune response to Innocell | Baseline to 30 days post last dose of Innocell
  Determined by > 1.5x over baseline via T-cell activation assay
Immunogenicity of Innocell Vaccine | Baseline to 30 days post last dose of Innocell
  Correlation of % cancer cells in Innocell vaccine to immune response
Clinical response | Baseline to 30 days post last dose of Innocell, with long-term FU every 3 months x 1 year
  Assessed by RECIST criteria v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- City of Hope, Duarte, California, United States